CLINICAL TRIAL: NCT00588809
Title: A Phase 2 Study of AZD6244 in Relapsed or Refractory AML
Brief Title: Selumetinib in Treating Patients With Recurrent or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00250; 15455B; N01CM62209 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Results first posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2013-02

CONDITIONS: Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Promyelocytic Leukemia (M3); Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute | interventions — AZD 6244

ARMS (1):
- Treatment (selumetinib) (Experimental): Patients receive selumetinib PO BID on days 1 -28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: selumetinib

INTERVENTIONS:
Drug: selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244

SUMMARY:
This phase II clinical trial is studying how well selumetinib works in treating patients with recurrent or refractory acute myeloid leukemia. Selumetinib may stop the growth of cancer by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (includes complete response-CR, complete response with incomplete count recovery CRi, partial response-PR, and minor response-MR) to AZD6244 (selumetinib).

SECONDARY OBJECTIVES:

I. To determine the effects of AZD6244 in AML samples on p-ERK and evaluate the potential utility of p-ERK inhibition as a surrogate marker of biologic activity.

II. To correlate the effects of AZD6244 with the presence (or absence) of mutated RAS or FLT-3 at baseline.

III. To assess the safety profile of AZD6244 in patients with AML.

OUTLINE:

Patients receive selumetinib orally (PO) twice daily (BID) on days 1 -28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Relapsed or refractory acute myeloid leukemia (AML)
  * Secondary AML including AML arising from antecedent hematologic diseases (e.g., myelodysplastic syndrome, myeloproliferative disorders, or therapy-related AML)
* Elderly patients ≥ 60 years of age, previously untreated, and who are not candidates for or have refused standard chemotherapy are eligible for this trial
* Patients with relapsed acute promyelocytic leukemia (APL) who are FLT3+ and have failed both tretinoin and arsenic therapy are eligible for this trial
* No known active CNS disease
* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Total bilirubin ≤ 2 mg/dL (unless due to disease, hemolysis, or Gilbert disease)

  * In patients with associated hemolysis or Gilbert disease, a bilirubin of > 2 mg/dL is allowed as a result of predominantly unconjugated hyperbilirubinemia
* AST/ALT < 3 times upper limit of normal
* Creatinine < 2 mg/dL
* Baseline pulse oximetry > 92%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 4 weeks (16 week for males) after completion of study treatment
* Recovered from prior therapy
* At least 2 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy

  * Hydroxyurea may be administered for the first 7 days of therapy in patients with rapidly rising white count (WBC > 20 K/μL)
* At least 4 weeks since prior investigational agents
* No prior MEK inhibitors
* No concurrent medication that can prolong the QT interval
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biological composition to AZD6244 or its excipient Captisol®
* QTc interval > 450 msecs or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, or family history of long QT interval syndrome), including New York Heart Association class III or IV heart failure
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness or social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-12; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Result] Jain N, Curran E, Iyengar NM, Diaz-Flores E, Kunnavakkam R, Popplewell L, Kirschbaum MH, Karrison T, Erba HP, Green M, Poire X, Koval G, Shannon K, Reddy PL, Joseph L, Atallah EL, Dy P, Thomas SP, Smith SE, Doyle LA, Stadler WM, Larson RA, Stock W, Odenike O. Phase II study of the oral MEK inhibitor selumetinib in advanced acute myelogenous leukemia: a University of Chicago phase II consortium trial. Clin Cancer Res. 2014 Jan 15;20(2):490-8. doi: 10.1158/1078-0432.CCR-13-1311. Epub 2013 Oct 31. PMID 24178622

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A Simon, optimal two-stage design was employed for subjects without FLT3 ITD mutations. The study also included a second cohort of subjects with FLT3 ITD mutations.
Groups:
- Selumetinib: Patients receive selumetinib PO BID on days 1 -28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  selumetinib: Given PO
Period: Overall Study
Arm/Group | Selumetinib
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Selumetinib
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 69 [26 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Response Rate for Subjects Without FLT3 ITD Mutation
Description: Responses were defined using standard criteria developed by an International Working Group.
  [Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, et al. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol 2003;21:4642-9.]
  In this primary outcome, we report the proportion of subjects without FLT3 ITD mutation that experienced a complete response (CR), partial response (PR), minor response (MR), or unconfirmed minor response (uMR).
Time Frame: Up to 52 weeks
Population: Analysis only includes subjects without FLT3 ITD mutation.
Measure: Number; unit: percentage of participants
Arm/Group | Selumetinib
Number analyzed (Participants) | 36
percentage of participants | 16.67

2. Secondary Outcome: Proportion of Subjects With Baseline p-ERK Activation
Description: Proportion of subjects with baseline p-ERK activation
Time Frame: baseline (0 weeks)
Population: The analysis includes the 20 patients with samples available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Selumetinib
Number analyzed (Participants) | 20
percentage of participants | 85

3. Secondary Outcome: Proportion of Subjects With NRAS Mutation
Description: Proportion of Subjects With NRAS Mutation
Time Frame: baseline (0 weeks)
Population: The analysis includes the 41 patients with samples available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Selumetinib
Number analyzed (Participants) | 41
percentage of participants | 7

4. Secondary Outcome: Proportion of Subjects With KRAS Mutation
Description: Proportion of subjects with KRAS mutation
Time Frame: baseline (0 weeks)
Population: The analysis includes the 41 patients with samples available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Selumetinib
Number analyzed (Participants) | 41
percentage of participants | 2

5. Secondary Outcome: Proportion of Subjects With FLT3 ITD Mutation
Description: Proportion of subjects with FLT3 ITD mutation
Time Frame: baseline (0 weeks)
Population: FLT3 ITD mutation status was not available for one patient.
Measure: Number; unit: percentage of participants
Arm/Group | Selumetinib
Number analyzed (Participants) | 46
percentage of participants | 22

6. Secondary Outcome: Proportion of Subjects With KIT Mutation
Description: Proportion of subjects with KIT mutation
Time Frame: baseline (0 weeks)
Population: The analysis includes the 41 patients with samples available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Selumetinib
Number analyzed (Participants) | 41
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Selumetinib
Serious Adverse Events (participants affected / at risk) | 38/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selumetinib (N=47)
Anemia (Blood and lymphatic system disorders) | 2 — A disorder characterized by an reduction in the amount of hemoglobin in 100 ml of blood.
Febrile neutropenia (Blood and lymphatic system disorders) | 8 — A disorder characterized by an ANC <1000/mm3 and a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour
Ventricular tachycardia (Cardiac disorders) | 1 — A disorder characterized by a dysrhythmia with a heart rate greater than 100 beats per minute that originates distal to the bundle of His.
Diarrhea (Gastrointestinal disorders) | 2 — A disorder characterized by frequent and watery bowel movements.
Dry mouth (Gastrointestinal disorders) | 1 — A disorder characterized by reduced salivary flow in the oral cavity.
Mucositis oral (Gastrointestinal disorders) | 2 — A disorder characterized by inflammation of the oral mucosal.
Nausea (Gastrointestinal disorders) | 2 — A disorder characterized by a queasy sensation and/or the urge to vomit.
Vomiting (Gastrointestinal disorders) | 3 — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
Death NOS (General disorders) | 10 — A cessation of life that cannot be attributed to a CTCAE term associated with Grade 5.
Fatigue (General disorders) | 3 — A disorder characterized by a state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities.
Fever (General disorders) | 2 — A disorder characterized by elevation of the body's temperature above the upper limit of normal.
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Blood (Infections and infestations) | 4
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Lung (pneumonia) (Infections and infestations) | 3
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Rectum (Infections and infestations) | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Salivary gland (Infections and infestations) | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Skin (cellulitis) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Blood (Infections and infestations) | 2
Infections and infestations - Other (Infections and infestations) | 11
Lung infection (Infections and infestations) | 3 — A disorder characterized by an infectious process involving the lungs.
peritonsillar abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1 — A disorder characterized by inflammation of the throat.
Sepsis (Infections and infestations) | 1 — A disorder characterized by the presence of pathogenic microorganisms in the blood stream that cause a rapidly progressing systemic reaction that may lead to shock.
Upper respiratory infection (Infections and infestations) | 1 — A disorder characterized by an infectious process involving the upper respiratory tract (nose, paranasal sinuses, pharynx, larynx, or trachea).
Urinary tract infection (Infections and infestations) | 1 — A disorder characterized by an infectious process involving the urinary tract, most commonly the bladder and the urethra.
Alanine aminotransferase increased (Investigations) | 1 — A finding based on laboratory test results that indicate an increase in the level of alanine aminotransferase (ALT or SGPT) in the blood specimen.
Creatinine increased (Investigations) | 1 — A finding based on laboratory test results that indicate increased levels of creatinine in a biological specimen.
Neutrophil count decreased (Investigations) | 1 — A finding based on laboratory test results that indicate a decrease in number of neutrophils in a blood specimen.
Platelet count decreased (Investigations) | 3 — A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen.
White blood cell decreased (Investigations) | 1 — A finding based on laboratory test results that indicate an decrease in number of white blood cells in a blood specimen.
Acidosis (Metabolism and nutrition disorders) | 1 — A disorder characterized by abnormally high acidity (high hydrogen-ion concentration) of the blood and other body tissues.
Anorexia (Metabolism and nutrition disorders) | 1 — A disorder characterized by a loss of appetite.
Dehydration (Metabolism and nutrition disorders) | 5 — A disorder characterized by excessive loss of water from the body. It is usually caused by severe diarrhea, vomiting or diaphoresis.
Hyperuricemia (Metabolism and nutrition disorders) | 1 — A disorder characterized by laboratory test results that indicate an elevation in the concentration of uric acid.
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 — A disorder characterized by laboratory test results that indicate a low concentration of albumin in the blood.
Hypokalemia (Metabolism and nutrition disorders) | 1 — A disorder characterized by laboratory test results that indicate a low concentration of potassium in the blood.
Hyponatremia (Metabolism and nutrition disorders) | 1 — A disorder characterized by laboratory test results that indicate a low concentration of sodium in the blood.
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 — A disorder characterized by a reduction in the strength of the lower limb muscles.
Dizziness (Nervous system disorders) | 2 — A disorder characterized by a disturbing sensation of lightheadedness, unsteadiness, giddiness, spinning or rocking.
Dysphasia (Nervous system disorders) | 1 — A disorder characterized by impairment of verbal communication skills, often resulting from brain damage.
Intracranial hemorrhage (Nervous system disorders) | 4 — A disorder characterized by bleeding from the cranium.
Psychosis (Psychiatric disorders) | 1 — A disorder characterized by personality change, impaired functioning, and loss of touch with reality. It may be a manifestation of schizophrenia, bipolar disorder or brain tumor.
Urine discoloration (Renal and urinary disorders) | 1 — A disorder characterized by a change in the color of the urine.
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 — A disorder characterized by bleeding from the bronchial wall and/or lung parenchyma.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 — A disorder characterized by an uncomfortable sensation of difficulty breathing.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 — A disorder characterized by bleeding from the nose.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 — A disorder characterized by a decrease in the level of oxygen in the body.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 — A disorder characterized by inflammation focally or diffusely affecting the lung parenchyma.
Hypotension (Vascular disorders) | 3 — A disorder characterized by a blood pressure that is below the normal expected for an individual in a given environment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selumetinib (N=47)
Anemia (Blood and lymphatic system disorders) | 24 — A disorder characterized by an reduction in the amount of hemoglobin in 100 ml of blood.
Febrile neutropenia (Blood and lymphatic system disorders) | 3 — A disorder characterized by an ANC <1000/mm3 and a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour
Atrial fibrillation (Cardiac disorders) | 3 — A disorder characterized by a dysrhythmia without discernible P waves and an irregular ventricular response due to multiple reentry circuits. The rhythm disturbance originates above the ventricles.
Paroxysmal atrial tachycardia (Cardiac disorders) | 4 — A disorder characterized by a dysrhythmia with abrupt onset and sudden termination of atrial contractions with a rate of 150-250 beats per minute. The rhythm disturbance originates in the atria.
Sinus tachycardia (Cardiac disorders) | 13 — A disorder characterized by a dysrhythmia with a heart rate greater than 100 beats per minute that originates in the sinus node.
Abdominal distension (Gastrointestinal disorders) | 7 — A disorder characterized by swelling of the abdomen.
Abdominal pain (Gastrointestinal disorders) | 13 — A disorder characterized by a sensation of marked discomfort in the abdominal region.
Constipation (Gastrointestinal disorders) | 4 — A disorder characterized by irregular and infrequent or difficult evacuation of the bowels.
Diarrhea (Gastrointestinal disorders) | 29 — A disorder characterized by frequent and watery bowel movements.
Dry mouth (Gastrointestinal disorders) | 6 — A disorder characterized by reduced salivary flow in the oral cavity.
Dyspepsia (Gastrointestinal disorders) | 3 — A disorder characterized by an uncomfortable, often painful feeling in the stomach, resulting from impaired digestion. Symptoms include burning stomach, bloating, heartburn, nausea and vomiting.
Hemorrhoids (Gastrointestinal disorders) | 4 — A disorder characterized by the presence of dilated veins in the rectum and surrounding area.
Mucositis oral (Gastrointestinal disorders) | 9 — A disorder characterized by inflammation of the oral mucosal.
Nausea (Gastrointestinal disorders) | 24 — A disorder characterized by a queasy sensation and/or the urge to vomit.
Oral hemorrhage (Gastrointestinal disorders) | 5 — A disorder characterized by bleeding from the mouth.
Vomiting (Gastrointestinal disorders) | 15 — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
Chills (General disorders) | 16 — A disorder characterized by a sensation of cold that often marks a physiologic response to sweating after a fever.
Edema limbs (General disorders) | 21 — A disorder characterized by swelling due to excessive fluid accumulation in the upper or lower extremities.
Fatigue (General disorders) | 32 — A disorder characterized by a state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities.
Fever (General disorders) | 21 — A disorder characterized by elevation of the body's temperature above the upper limit of normal.
Non-cardiac chest pain (General disorders) | 7 — A disorder characterized by discomfort in the chest unrelated to a heart disorder.
Pain (General disorders) | 6 — A disorder characterized by the sensation of marked discomfort, distress or agony.
Allergic reaction (Immune system disorders) | 5 — A disorder characterized by an adverse local or general response from exposure to an allergen.
Infections and infestations - Other (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 3 — A disorder characterized by an infectious process involving the urinary tract, most commonly the bladder and the urethra.
Bruising (Injury, poisoning and procedural complications) | 3 — A finding of injury of the soft tissues or bone characterized by leakage of blood into surrounding tissues.
Alanine aminotransferase increased (Investigations) | 16 — A finding based on laboratory test results that indicate an increase in the level of alanine aminotransferase (ALT or SGPT) in the blood specimen.
Alkaline phosphatase increased (Investigations) | 7 — A finding based on laboratory test results that indicate an increase in the level of alkaline phosphatase in a blood specimen.
Aspartate aminotransferase increased (Investigations) | 19 — A finding based on laboratory test results that indicate an increase in the level of aspartate aminotransferase (AST or SGOT) in a blood specimen.
Blood bilirubin increased (Investigations) | 5 — A finding based on laboratory test results that indicate an abnormally high level of bilirubin in the blood. Excess bilirubin is associated with jaundice.
Creatinine increased (Investigations) | 7 — A finding based on laboratory test results that indicate increased levels of creatinine in a biological specimen.
Lymphocyte count decreased (Investigations) | 8 — A finding based on laboratory test results that indicate a decrease in number of lymphocytes in a blood specimen.
Neutrophil count decreased (Investigations) | 20 — A finding based on laboratory test results that indicate a decrease in number of neutrophils in a blood specimen.
Platelet count decreased (Investigations) | 24 — A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen.
Weight loss (Investigations) | 3 — A finding characterized by a decrease in overall body weight; for pediatrics, less than the baseline growth curve.
White blood cell decreased (Investigations) | 13 — A finding based on laboratory test results that indicate an decrease in number of white blood cells in a blood specimen.
Acidosis (Metabolism and nutrition disorders) | 5 — A disorder characterized by abnormally high acidity (high hydrogen-ion concentration) of the blood and other body tissues.
Anorexia (Metabolism and nutrition disorders) | 19 — A disorder characterized by a loss of appetite.
Dehydration (Metabolism and nutrition disorders) | 4 — A disorder characterized by excessive loss of water from the body. It is usually caused by severe diarrhea, vomiting or diaphoresis.
Hyperglycemia (Metabolism and nutrition disorders) | 17 — A disorder characterized by laboratory test results that indicate an elevation in the concentration of blood sugar. It is usually an indication of diabetes mellitus or glucose intolerance.
Hyperuricemia (Metabolism and nutrition disorders) | 3 — A disorder characterized by laboratory test results that indicate an elevation in the concentration of uric acid.
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 — A disorder characterized by laboratory test results that indicate a low concentration of albumin in the blood.
Hypocalcemia (Metabolism and nutrition disorders) | 13 — A disorder characterized by laboratory test results that indicate a low concentration of calcium (corrected for albumin) in the blood.
Hypoglycemia (Metabolism and nutrition disorders) | 3 — A disorder characterized by laboratory test results that indicate a low concentration of glucose in the blood.
Hypokalemia (Metabolism and nutrition disorders) | 12 — A disorder characterized by laboratory test results that indicate a low concentration of potassium in the blood.
Hypomagnesemia (Metabolism and nutrition disorders) | 9 — A disorder characterized by laboratory test results that indicate a low concentration of magnesium in the blood.
Hyponatremia (Metabolism and nutrition disorders) | 15 — A disorder characterized by laboratory test results that indicate a low concentration of sodium in the blood.
Hypophosphatemia (Metabolism and nutrition disorders) | 5 — A disorder characterized by laboratory test results that indicate a low concentration of phosphates in the blood.
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 — A disorder characterized by a sensation of marked discomfort in a joint.
Back pain (Musculoskeletal and connective tissue disorders) | 9 — A disorder characterized by marked discomfort sensation in the back region.
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 — A disorder characterized by a reduction in the strength of muscles in multiple anatomic sites.
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 — A disorder characterized by a reduction in the strength of the lower limb muscles.
Dizziness (Nervous system disorders) | 10 — A disorder characterized by a disturbing sensation of lightheadedness, unsteadiness, giddiness, spinning or rocking.
Headache (Nervous system disorders) | 12 — A disorder characterized by a sensation of marked discomfort in various parts of the head, not confined to the area of distribution of any nerve.
Confusion (Psychiatric disorders) | 4 — A disorder characterized by a lack of clear and orderly thought and behavior.
Depression (Psychiatric disorders) | 4 — A disorder characterized by melancholic feelings of grief or unhappiness.
Proteinuria (Renal and urinary disorders) | 4 — A disorder characterized by laboratory test results that indicate the presence of excessive protein in the urine. It is predominantly albumin, but also globulin.
Urinary retention (Renal and urinary disorders) | 3 — A disorder characterized by accumulation of urine within the bladder because of the inability to urinate.
Cough (Respiratory, thoracic and mediastinal disorders) | 18 — A disorder characterized by sudden, often repetitive, spasmodic contraction of the thoracic cavity, resulting in violent release of air from the lungs and usually accompanied by a distinctive sound.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 — A disorder characterized by an uncomfortable sensation of difficulty breathing.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 — A disorder characterized by bleeding from the nose.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 — A disorder characterized by a decrease in the level of oxygen in the body.
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 — A disorder characterized by marked discomfort sensation in the pharyngolaryngeal region.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 — A disorder characterized by an increase in amounts of fluid within the pleural cavity. Symptoms include shortness of breath, cough and marked chest discomfort.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 — A disorder characterized by inflammation focally or diffusely affecting the lung parenchyma.
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 — A disorder characterized by flaky and dull skin; the pores are generally fine, the texture is a papery thin texture.
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 — A disorder characterized by excessive perspiration.
Purpura (Skin and subcutaneous tissue disorders) | 4 — A disorder characterized by hemorrhagic areas of the skin and mucous membrane. Newer lesions appear reddish in color. Older lesions are usually a darker purple color and eventually become a brownish-yellow color.
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 — A disorder characterized by the presence of macules (flat) and papules (elevated). Also known as morbillform rash.
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 9 — A disorder characterized by a pathological increase in blood pressure; a repeatedly elevation in the blood pressure exceeding 140 over 90 mm Hg.
Hypotension (Vascular disorders) | 7 — A disorder characterized by a blood pressure that is below the normal expected for an individual in a given environment.
Vascular disorders - Other (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less